CLINICAL TRIAL: NCT05562167
Title: The Inorganic Nitrate and eXercise Performance in Heart Failure (iNIX-HF) -a Phase II Clinical Trial
Brief Title: The Inorganic Nitrate and eXercise Performance in Heart Failure (iNIX-HF)
Acronym: iNIX-HF
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202204141
Record Dates: First submitted 2022-09-21; First posted 2022-09-30 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — potassium nitrate

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, parallel arm design
Who Masked: Participant, Investigator
Masking Description: Double blind, placebo controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Potassium Nitrate (KNO3) treatment arm (Experimental): 10 mmol of KNO3 via a single gel capsule to be consumed orally once per day for 6 weeks.
  Interventions: Drug: KNO3
- Placebo-controlled arm (Placebo Comparator): 10 mmol of placebo via a single gel capsule to be consumed orally once per day for 6 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KNO3 — 10 mmol of KNO3 via a single gel capsule to be consumed orally once per day for 6 weeks.
  Other Names: Potassium nitrate
  Arms: Potassium Nitrate (KNO3) treatment arm
Drug: Placebo — 10 mmol of placebo via a single gel capsule to be consumed orally once per day for 6 weeks.
  Arms: Placebo-controlled arm

SUMMARY:
The goals of this project are to determine the effectiveness of acute (2 hours after a single dose) and chronic (after 6 weeks of once-a-day dosing) KNO3 treatment (10mmol) vs. placebo on quadriceps muscle power and on aerobic exercise performance (V̇O2peak) in patients with HFrEF (left ventricular ejection fraction <45%). The investigators hypothesize that both acute and chronic dosing of 10mmol of KNO3 will improve exercise performance in HFrEF. To test this hypothesis, the investors will perform a randomized, double-blind, placebo-controlled, parallel-arm design study.

DETAILED DESCRIPTION:
Visit 1 Screening/Phenotyping Day.

1. Consent: All study procedures will be reviewed with the participants before the investigators obtain written informed consent. Consent includes giving permission for the investigators to review their medical records.
2. Blood Samples: Participants will report to the Clinical Translational Research Unit (CTRU) at Washington University Medical Center after an overnight (10-12 hour) fast. An intravenous catheter will be placed to facilitate blood sampling 5 times during the visit. The first blood sample (time 0) will be for screening/phenotyping laboratories: NT-proBNP, chemistries (including K+), glucose, and creatinine (for estimation of glomerular filtration rate).
3. Urine Pregnancy Test: Women of child-bearing age will have a urine pregnancy test.
4. Physical Exam: Participants will have a brief history and physical examination. Heart rate (HR) and blood pressure (BP) will be taken.
5. Resting Echocardiogram with contrast: Participants will also undergo a standard 2D Doppler, tissue Doppler and strain imaging echocardiography to quantify left ventricular structure and function.
6. Questionnaires: Participants will complete a medical history form, the Kansas City Cardiomyopathy Questionnaire (KCCQ), and Minnesota Living with Heart Failure Questionnaire (MLHFQ).
7. NYHA classification will be determined.
8. Blood Pressure and Heart Rate: BP and HR will be measured at time 0 and hourly for 4 hours.
9. Breath Nitric Oxide: Participants will exhale into a tube attached to a portable electrochemical analyzer (NIOX VERO, Aerocrine Inc., Morrisville, NC) following the American Thoracic Society/European Respiratory Society guidelines at time 0 and hourly for 4 hours.
10. Blood sampling for NO3- and NO2-: Participants will have blood drawn (20mL or about 1.5 tbsp) through their previously placed intravenous catheter at time 0 and hourly for 4 hours.
11. Exercise Test - Maximal Muscle Power: After 2 hours, knee extensor muscle power will be determined using a Biodex isokinetic dynamometer (Biodex Medical Systems, Shirley, NY).
12. Exercise Test - Aerobic Capacity: After 10 min of recovery from the muscle power testing, peak oxygen consumption (V̇O2peak) will be determined with an incremental treadmill exercise test to volitional fatigue.
13. Randomization: Participants will be randomized to the KNO3 or placebo arm in a double-blind fashion, stratified by sex and ischemic/nonischemic status.
14. Participants will be instructed to take the medication every day at the same time of the AM. Participants will be instructed to take the medication with food.

    Visit 2: Acute Dose Study Day
15. Baseline blood K+ and eGFR levels. As with Visit 1, participants will report to the CTRU fasted (and not having used mouthwash for 24 hours) and have a physical exam and blood drawn for creatinine and K+.
16. Ingestion of a gelatin capsule containing either 10 mmol KNO3 or placebo, per the randomization scheme.
17. HR, BP, plasma NO3- and NO2- , and breath NO: As in Visit 1, HR, BP, plasma NO3- and NO2- , and breath NO will be measured at time 0 (prior to ingestion of a single gelatin capsule) and thereafter hourly for 4 h after the participant ingests a single gelatin capsule containing either 10 mmol KNO3 or placebo, per the randomization scheme.
18. Exercise Test - Maximal Muscle Power: After 2 hours, knee extensor muscle power will be determined using a Biodex isokinetic dynamometer.
19. Exercise Test - Aerobic Capacity: After 10 min of recovery from the muscle power testing, peak oxygen consumption (V̇O2peak) will be determined with an incremental treadmill exercise test to volitional fatigue.
20. Questionnaires: Participants will complete a medical history form, the Kansas City Cardiomyopathy Questionnaire (KCCQ), and Minnesota Living with Heart Failure Questionnaire (MLHFQ).
21. Intervention: After completion of Visit 2, participants will be given a 6-week course of 10 mmol KNO3 or placebo (such that the participants will be given the same medication (nitrate or placebo) that they were given in the Acute Dose Study), one capsule for each day, to be taken p.o.. Participants will be instructed to not use mouthwash before ingesting the study capsules and to not change their diet or level of physical activity during the study (in particular, to not begin or cease an exercise program while enrolled in the study).

    Visit 3: 6-Week Dose
22. Procedures: The procedures for this visit will be identical to those described for Visit 2.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of heart failure with reduced ejection fraction; New York Heart Association (NYHA) Class II-III; Ejection fraction less than 45% as determined on an imaging study within 3 months of enrollment.
* Stable medical therapy, defined by no addition or removal (or change of more than 100 percent) of the following: beta-adrenergic blockade and angiotensin converting enzyme (ACE) inhibitors or angiotensin receptor blocker (ARB or aldosterone antagonists) or ARNI (ARB + sacubitril) for 60 days.

Exclusion Criteria:

* Vulnerable populations as defined by the U.S. Department of Health and Human Services; prisoners and children will be excluded from this study
* Pharmacologic, organic nitrate therapy within the last 3 months
* Major orthopedic, psychiatric, neurological, or other conditions that would hinder the ability to complete the exercise tests
* Estimated glomerular filtration rate less than 45 mL/min on screening clinical laboratories
* Systolic blood pressure less than 90mmHg or greater than 180mmHg at screening; Diastolic blood pressure less than 40mmHg or greater than 100mmHg at screening
* Previous adverse reaction to nitrate necessitating withdrawal of therapy; Treatment with phosphodiesterase inhibitors within the last 3 months (patient must also be willing to not take them for the duration of the trial)
* Ejection fraction greater than or equal to 45%
* Primary hypertrophic cardiomyopathy; Infiltrative cardiomyopathy (e.g., amyloid); Active myocarditis; Complex congenital heart disease;
* Active collagen vascular disease;
* Percutaneous coronary intervention, new bi-ventricular pacing, or coronary artery bypass grafting within the past 3 months
* Valvular heart disease with severe regurgitation or stenosis of any valve
* Acute or chronic severe liver disease as evidenced by encephalopathy or variceal bleeding
* Terminal disease (other than heart failure) with expected survival less than 1 y
* Enrollment in another therapeutic trial during the period of the study
* Pregnant women; Postmenopausal women taking exogenous estrogen replacement therapy
* Patients requiring exogenous oxygen at rest or during exercise
* Patients with active angina or ischemia due to epicardial coronary disease
* Patients taking xanthine oxidase inhibitors will be excluded
* Individuals taking proton pump inhibitors, antacids will be asked to hold these medications for the duration of the study if approved by his/her physician.

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-03-31 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
VO2 Peak Testing | Determined at Visit 1, Visit 2, and Visit 3, which will be scheduled throughout 8 weeks.
  peak oxygen consumption during treadmill exercise
Maximal muscle power | Determined at Visit 1, Visit 2, and Visit 3, which will be scheduled throughout 8 weeks.
  assessment of quadriceps power

SECONDARY OUTCOMES:
MLHFQ questionnaire | Determined at Visit 1, Visit 2, and Visit 3, which will be scheduled throughout 8 weeks.
  Minnesota Living with Heart Failure Questionnaire
KCCQ questionnaire | Determined at Visit 1, Visit 2, and Visit 3, which will be scheduled throughout 8 weeks.
  Kansas City Cardiomyopathy Questionnaire
Maximal muscle velocity | Determined at Visit 1, Visit 2, and Visit 3, which will be scheduled throughout 8 weeks.
  assessment of quadriceps velocity
Maximal exercise time on treadmill | Determined at Visit 1, Visit 2, and Visit 3, which will be scheduled throughout 8 weeks.
  Maximum time spent on treadmill during the VO2 peak test
Plasma nitrate and nitrite | Determined at Visit 1, Visit 2, and Visit 3, which will be scheduled throughout 8 weeks.
  concentrations of nitrate and nitrite in the blood
Breath nitric oxide (NO) level | Determined at Visit 1, Visit 2, and Visit 3, which will be scheduled throughout 8 weeks.
  breath NO level

CONTACTS AND LOCATIONS:
Overall Officials: Linda R Peterson, MD, Principal Investigator — Washington University School of Medicine; Lauren K Park, PhD, Study Director — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States